CLINICAL TRIAL: NCT02752022
Title: Monitoring Levels of Tobacco-specific Nitrosamines, DNA Adducts, Stress Hormones and DNA Methylation During the Transition From Cigarette Smoking to Electronic Cigarette Use: a Prospective Observational Study
Brief Title: Monitoring the Transition From Smoking to E-cigarettes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 16.0070
Record Dates: First submitted 2016-04-13; First posted 2016-04-26 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Smoking
Keywords: e-cigarettes; nitrosamines; smoking cessation
MeSH Terms: conditions — Smoking; Vaping; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, bucal swab, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heavy smokers: Heavy smokers (continuous smoking of >10 cigarettes per day) for at least 6 months who will give up smoking and switch to nicotine containing e-cigarettes for 28 days to help them quit smoking.

SUMMARY:
Electronic cigarettes (e-cigarettes) have proved very popular and a meteoric rise in their usage is currently under way. People purchase them as an aid to giving up smoking, to reduce cigarette consumption, to minimise withdrawal symptoms in occupational environments that ban smoking, and in order to continue smoking with decreased health risks. Although the safety and impact on health of electronic cigarettes, especially after long-term use, has not been evaluated, they are generally considered to be far safer alternatives to cigarette smoke. Electronic cigarettes do not generate polycyclic aromatic hydrocarbons, a potent class of carcinogenic chemicals generated during the combustion of tobacco and making important contribution to the cigarette-induced cancer. However, carcinogenic tobacco-specific nitrosamines have been encountered in e-cigarettes being detected in some nicotine cartridges as contaminants, albeit at very low concentrations in comparison with tobacco smoke. Consequently, it is imperative to ascertain the toxicity risk (if any) of consuming nicotine intake through electronic cigarettes. This European Commission funded study will monitor levels of carcinogenic tobacco-specific nitrosamines in urine of heavy smokers who give up smoking and completely transition to e-cigarette use for a period of 4 weeks. Levels of other compounds which are known to be associated with smoking toxicity, such as DNA adducts and DNA methylation, will also be monitored in biological fluids of these subjects. Finally, cigarette craving, mood, anxiety, social anxiety, well-being status and stress hormones will be measured in smokers transitioning to e-cigarettes for 4 weeks to assess the psychological effect of the transition. The results from the study will provide important information on the safety and effectiveness of e-cigarettes for smoking cessation which investigators anticipate to drive policy.

DETAILED DESCRIPTION:
Established smokers will completely stop smoking for 4 weeks and instead transition to nicotine use through an electronic cigarette as required. They will be free to purchase the e-cigarette and e-liquid/cartridges of their own choice.

Eligible subjects will be asked to visit St George's Clinical Research Facility to provide the following samples. Blood, saliva and buccal cells to be collected on screening day. 24hr urine, blood, saliva and buccal cells will be collected at baseline and on days 3, 7, 21 and 28 after the first transition to e-cigarette use.

Moreover, subjects will be breathalysed with carbon monoxide (CO) oximeter and their urine analysed for anatabine to assess compliance to the study protocol (complete refrain of use of tobacco cigarettes for 4 weeks while they use e-cigarettes).

Subjects will be monitored for craving, mood, social anxiety, sleep profile and quality of life on every visit to St George's Clinical Research Facility (quality of life will be assessed only at baseline and day 28 of e-cigarette use). The subjects will be followed up with a telephone call 6 and 12 months after the end of the e-cigarette intervention to monitor their smoking/e-cigarette use behaviour and participants craving, mood, social anxiety, sleep profile and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Heavy smokers (continuous smoking of >10 cigarettes per day) for at least 6 months who are willing to give up smoking and switch to nicotine containing e-cigarettes to help them quit smoking.
2. Males and females aged 18-65 years
3. Subjects must be willing and able to give informed consent
4. Subjects must have understanding of English sufficient that they are able to read and understand the participant information sheet and the informed consent form
5. Subjects in the opinion of the Investigator are healthy on the basis of medical history questionnaire and vital signs
6. Subjects who will purchase their e-cigarettes kits, e-liquid and/or cartridges from a pharmacy, leading super market, established newsagent chain)

Exclusion Criteria:

1. Severe psychosis, Bipolar Affective Disorder I, prostate cancer, Cushing's syndrome, severe depression with suicidal ideation and intention, brain trauma or other severe neurological disorders (e.g. pan-hypopituitarism) or taking antidepressants, anxiolytics antipsychotics
2. Pregnant females and lactating mothers
3. History of substance abuse and alcoholism
4. History of cardiovascular disease (heart disease, angina, heart attacks, high blood pressure, heart surgery) in the last 6 months.
5. Self-declared smokers with low or non-detectable CO readings in their breath when tested with the oxymeter will be excluded from further being studied
6. Smokers who are undergoing alternative Nicotine Replacement Therapy (NRT)/pharmacological treatment for smoking cessation (i.e. nicotine patches, nicotine gum, Champix, bupropion)
7. Any other condition that in the judgement of the investigator would preclude participation
8. Smokers who are unwilling to refrain from smoking for 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heavy smokers (continuous smoking of >10 cigarettes per day) for at least 6 months who are willing to give up smoking and switch to nicotine containing e-cigarettes to help them quit smoking
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Change of levels of DNA adducts analysed by high resolution liquid chromatography | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Change of levels of tobacco specific nitrosamines analysed by high resolution liquid chromatography | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Change of levels of stress hormones analysed by ELISA | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Change of levels of DNA methylation analysed by high pressure liquid chromatography-UV | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes

SECONDARY OUTCOMES:
Change of measures of withdrawal symptoms severity measured by the Fagerstrom test | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Change of measures of craving analysed by Minnesota Nicotine Withdrawal Scale | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Change of measures of mood analysed by Mood and Physical Symptoms Scale (MPSS) | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Change of measures of anxiety analysed by State-Trait Anxiety Inventory | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Change of measures of social anxiety analysed by Liebovitz Social Anxiety Test | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Changes of measures of depression analysed by Beck Depression Inventory | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Changes of measures of sleep analysed by Pittsburg Sleep Index or Karolinska sleep questionaire | Screening, baseline and 3, 7, 21 and 28 days following transition to e-cigarettes
Changes of measure of quality of life analysed by the European Quality of Life Questionnaire (EuroQL-5D) | baseline and 28 days following transition to e-cigarettes
Changes in brain electrical activity measured by EEG | baseline and 21 days following transition to e-cigarettes

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Bailey, Principal Investigator — St George's, University of London
Locations (1):
- St George's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No